CLINICAL TRIAL: NCT03303508
Title: Detection Of Anti-Double Stranded Deoxyribonucleic Acid Antibodies In Autoimmune Rheumatic Diseases: Comparison Between Immunofluorescence And Enzyme Immunoassay
Brief Title: Measurement of Anti-dsDNA by Both CLIFT & ELISA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, SONagi, Detection of Anti-Double Stranded Deoxyribonucleic Acid Antibodies in Autoimmune Rheumatic Diseases, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLIFT & ELISA
Record Dates: First submitted 2017-09-27; First posted 2017-10-06 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-09

CONDITIONS: Antiphospholipid Syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Intervention Model Description: The study will include patients with suspected diagnosis of autoimmune rheumatic diseases referred to the Laboratory of Clinical Immunology, Clinical Pathology Department, Assiut University Hospital for anti-dsDNA test. Patients will be recruited into the study within period of one year.
  Also, apparently healthy subjects (at least 25 subjects; according to international method verification guidelines) will be included as a control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-ds DNA (Other): anti-ds DNA
  Interventions: Diagnostic Test: anti-ds DNA

INTERVENTIONS:
Diagnostic Test: anti-ds DNA — venous blood samples
  Other Names: venous blood samples

SUMMARY:
detection of anti-ds DNA in patients with rheumatic diseases by two methodes : immunofluorescence & ELISA

DETAILED DESCRIPTION:
Autoimmune rheumatic diseases are autoimmune disorders presented with joint and muscles manifestations. However, other organs may be involved at a varying degree in different conditions. They are also called connective tissue diseases (CTDs) or collagen diseases. They include systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), Sjiogren's syndrome (SjS), systemic sclerosis, polymyositis and dermatomyositis and mixed connective tissue disease (Peakman and Vergani, 2009).

Autoimmune rheumatic diseases are characterized by presence of antinuclear antibodies (ANA). These antibodies are involved in the disease pathogenesis, and their presence in patients' sera constitutes one of the criteria used (together with the clinical manifestations) for disease diagnosis (Stevens, 2010). ANA include autoantibodies to extractable nuclear antigens and autoantibodies to histones and deoxyribonucleic acid (DNA).

Anti-DNA antibodies include those against single and double stranded DNA (ssDNA and dsDNA, respectively). Anti-dsDNA antibodies are recognized as diagnostic markers of SLE and as indicators of SLE disease activity, especially in lupus nephritis (Zigon et al., 2011).However, high anti-dsDNA levels are found only in 50-70% of SLE patients. So, negative anti-dsDNA test does not exclude SLE Also, anti-dsDNA antibodies can be detected in other autoimmune diseases such as RA and SjS, as well as in healthy blood donors (Zigon et al., 2011).The significance of anti-dsDNA in SLE diagnosis and in monitoring SLE disease activity has led to an increase in this test laboratory requests as well as in the number of commercially available kits (Chiaro et al., 2011).

The kits that are used in detection and quantitation of anti-dsDNA antibodies include:

1. Radioimmunoassay methods developed according to Farr technique (FARR-RIA) (Wold et al., 1968). However, due to the use of radioactive element in the Farr assay, it is not widely used in the routine diagnostic laboratory work (Mahler and Fritzler, 2007).
2. Crithidia luciliae immunofluorescence test (CLIFT) developed by Aarden et al (1975) detects anti-dsDNA by indirect immunofluorescence using the hemoflagellate Crithidia luciliae which contains kinetoplast that contains a high concentration of native (dsDNA) DNA (Zigon et al., 2011). However, reading and interpretation of the immunoflourescence is subjective and depends on the experience and training of the laboratory personnel which could affects the test results (Chiaro et al., 2011).
3. Enzyme-linked immunosorbant assay (ELISA) is simple to perform, does not require highly trained operators and can be automated. Therefore, it is becoming the most widely used method (Kumar et al., 2009).With the increasing number of anti-dsDNA ELISA assays, the potential for variability in the diagnostic accuracies is enormous as different antigens, assay principles and cutoff determinations are employed (Chiaro et al., 2011). Anti- dsDNA ELISAs may give false-positive results due to binding of immune complexes to the pre-coat intermediates (Zigon et al., 2011).

In the Laboratory of Clinical Immunology, Assiut University Hospital, we shifted from manual ELISA kits to automated ELISA platform (Alegria system, Orgentec Diagnostika, Germany) and recently CLIFT was introduced in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients with suspected diagnosis of autoimmune rheumatic diseases referred to the Laboratory of Clinical Immunology, Clinical Pathology Department, Assiut University Hospital for anti-dsDNA test. Patients will be recruited into the study within period of one year.

Also, apparently healthy subjects (at least 25 subjects; according to international method verification guidelines) will be included as a control group

Exclusion Criteria:

* Subjects refused to be included in the study. Patients without a definite diagnosis of autoimmune rheumatic disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Comparison Between Immunofluorescence and Enzyme Immunoassay | one year
  Verfication of the anti-dsDNA examination methods used in the Laboratory of Clinical Immunology, Assiut University Hospital.

SECONDARY OUTCOMES:
Detection of Anti-Double Stranded Deoxyribonucleic Acid Antibodies in Autoimmune Rheumatic Diseases | one year
  Verfication of the anti-dsDNA examination

REFERENCES:
- [Background] Bai Y, Tong Y, Liu Y, Hu H. Self-dsDNA in the pathogenesis of systemic lupus erythematosus. Clin Exp Immunol. 2018 Jan;191(1):1-10. doi: 10.1111/cei.13041. Epub 2017 Sep 15. PMID 28836661